CLINICAL TRIAL: NCT04684160
Title: Comparison of Joint Awareness Between Fixed-bearing and Mobile-bearing Total Knee Arthroplasty Using Titanium-nitride Coated Posterior-stabilized Prostheses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUKorea MB
Record Dates: First submitted 2020-12-16; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis, Knee; Arthropathy of Knee; Joint Awareness
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed-bearing group (Active Comparator)
  Interventions: Device: Fixed-bearing TKA
- Mobile-bearing group (Experimental)
  Interventions: Device: Mobile-bearing TKA

INTERVENTIONS:
Device: Fixed-bearing TKA
  Arms: Fixed-bearing group
Device: Mobile-bearing TKA
  Arms: Mobile-bearing group

SUMMARY:
Comparison of postoperative patient's joint awareness as well as clinical and radiological outcomes between fixed- and mobile-bearing total knee arthroplasty of which the prosthesis is coated with Titanium-nitride.

DETAILED DESCRIPTION:
Despite numerous comparison studies between mobile- and fixed-bearing TKA as well as several comparison studies regarding clinical and radiological outcomes using titanium-nitride(TiN) prosthesis, there has been no study on postoperative joint awareness despite mobile- and fixed-bearing TKA using TiN prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee joint advanced osteoarthritis
* Age over 55 years old
* Scheduled to undergo primary total knee arthroplasty

Exclusion Criteria:

* Post-traumatic or inflammatory osteoarthritis
* Those who undertook previous ligamentous surgery
* Those who do not understand and give answers to a survey

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Forgotten joint score | Postoperative 3 years
  Questionnaire of evaluating how much the patients are aware of their operate joint during daily activities. The higher, the worse. Range: 0-100
Crepitus | Postoperative 3 years
  Any grating, crackling or popping sensation around knee when moving a joint

SECONDARY OUTCOMES:
Forgotten joint score | Postoperative 5 years
  Questionnaire of evaluating how much the patients are aware of their operate joint during daily activities. The higher, the worse. Range: 0-100
Crepitus | Postoperative 5 years
  Any grating, crackling or popping sensation around knee when moving a joint

OTHER OUTCOMES:
Change from baseline Knee Society Score (KSS) at 3 and 5 years | Preoperative and Postoperative 3, 5 years
  Patient-reported Outcome measure; The lower, the worse. Range: 0-200
Change from baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) at 3 and 5 years | Preoperative and Postoperative 3, 5 years
  Patient-reported Outcome measure; The higher, the worse. Range: 0-96
Central Sensitization Index (CSI) | Postoperative 3 years
  Questionnaire of evaluating how much the patients are sensitized on the pain. The higher, the worse. Range: 0-100
Central Sensitization Index (CSI) | Postoperative 5 years
  Questionnaire of evaluating how much the patients are sensitized on the pain. The higher, the worse. Range: 0-100
Radiological outcomes | Postoperative 3 years
  Measurements of radiological angles
Radiological outcomes | Postoperative 5 years
  Measurements of radiological angles

CONTACTS AND LOCATIONS:
Overall Officials: Yong In, M.D., Ph.D., Study Chair — Seoul St. Mary's Hospital
Locations (1):
- The Catholic University of Korea Seoul St Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No